CLINICAL TRIAL: NCT00885586
Title: Analgetic Effectiveness of Acupuncture When Compared to a Standardised Analgesic Regimen in the Treatment of Herpes Zoster Neuralgia
Brief Title: Acupuncture in Herpes Zoster Neuralgia (ACUZoster)
Acronym: ACUZoster
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dominik Irnich (Other)
Responsible Party: Sponsor-Investigator, Dominik Irnich, PD Dr. Dominik Irnich, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AcuZoster Effectiveness 2006
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Herpes Zoster; Postherpetic Neuralgia; Pain
Keywords: herpes zoster; neuropathic pain; acupuncture; randomised controlled trial; acute herpes zoster
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic; Pain; Neuralgia | interventions — Gabapentin; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sham-laser acupuncture (Sham Comparator): Sham laser acupuncture (c) is applied at equivalent points as needle acupuncture. Laser irradiation is faked.
  Interventions: Device: Sham-laser acupuncture
- gabapentine (Active Comparator): standard analgesic treatment
  Interventions: Drug: gabapentine
- Acupuncture (Active Comparator): Acupuncture treatment is semi-standardized, i.e. beside a scheme of basic points, individual points can be chosen according to the TCM diagnostic pattern.
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Device: Sham-laser acupuncture — Laser irradiation is faked, approaching a non-functioning laser pen.
  Arms: Sham-laser acupuncture
Drug: gabapentine — Patients in this arm are treated individually with gabapentine 900 mg/d - 3600 mg/d, according to the recommended scheme given by the manufacturer
  Arms: gabapentine
Procedure: Acupuncture — The needle acupuncture technique used in this trial is performed according the traditional way (TCM) using expendable needles.
  Arms: Acupuncture

SUMMARY:
Symptoms that herald herpes zoster include pruritus, dysesthesia and pain along the distribution of the involved dermatome. The most distressing symptom is typically pain and the most feared complication is postherpetic neuralgia (PHN), the persistence of pain long after rash healing. PHN is defined as pain persisting more than 3 months after the rash has healed. Both, the acute pain associated with herpes zoster and the chronic pain of PHN, have multiple adverse effects on health-related quality of life.

The primary objective of the trial presented is to investigate whether a 4 week semi-standardised acupuncture is non-inferior (first step) or superior (second step) to (a) the anticonvulsive drug gabapentin and (b) sham laser acupuncture in the treatment of pain associated with herpes zoster in addition to standardised analgesics. Secondary objectives include an assessment of the change of sensoric function, of long-term effectiveness, the occurrence of PHN and an evaluation of several pain specific questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acute HZ
* Pain intensity > 30 mm visual analog scale

Exclusion Criteria:

* Patients with insulin-dependent diabetes mellitus or other diseases influencing the peripheral sensibility (e.g., polyneuropathia, chronic pain syndromes, cutaneous irritations i.e. burns)
* Patients under age
* Uncompliance
* Pregnancy or lactation
* Surgery within the last 3 month
* Severe heart/lung/kidney disease
* Diseases influencing the quality of life
* Psychiatric diseases (e.g., depression, schizophrenia, dementia)
* Chronic intake of analgesics, neuroleptics, antidepressants, corticoids, alpha-agonists
* Acupuncture, transdermal electric neurostimulation or other Complementary and Alternative Medicine treatment within the last 4 weeks
* Contraindications according to the summary of product informations against analgesic treatment (i.e., metamizol, paracetamol, tramadol, morphine) or the investigational medicinal products (gabapentine, acupuncture needles)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-11; Primary Completion 2017-08-29 (Actual); Study Completion 2018-04-05 (Actual)

PRIMARY OUTCOMES:
Alteration of pain intensity after treatment | 5 weeks

SECONDARY OUTCOMES:
Quantitative sensory testing | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Multidisciplinary Pain Unit, University of Munich, Munich, Bavaria, Germany

REFERENCES:
- [Background] Fleckenstein J, Kramer S, Hoffrogge P, Thoma S, Lang PM, Lehmeyer L, Schober GM, Pfab F, Ring J, Weisenseel P, Schotten KJ, Mansmann U, Irnich D. Acupuncture in acute herpes zoster pain therapy (ACUZoster) - design and protocol of a randomised controlled trial. BMC Complement Altern Med. 2009 Aug 12;9:31. doi: 10.1186/1472-6882-9-31. PMID 19674449